CLINICAL TRIAL: NCT02099955
Title: Effects of Vitamin D Deficiency and Its Replacement on Pulmonary and Endocrine Function in Persons With SCI
Brief Title: Vitamin D Deficiency and Replacement on Pulmonary and Endocrine Function in SCI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Research Center Director, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAU-11-092
Record Dates: First submitted 2013-12-05; First posted 2014-03-31 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Spinal Cord Injury; Vitamin D Deficiency
Keywords: spinal cord injury; vitamin D deficiency; pulmonary function; metabolic diseases
MeSH Terms: conditions — Spinal Cord Injuries; Vitamin D Deficiency; Metabolic Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- Screening Study (No Intervention): To determine the prevalence and severity of vitamin D deficiency and glucose tolerance in persons with chronic SCI.
- Pulmonary Arm (Experimental): Vitamin D3 Supplementation and Pulmonary Function:
  1. To determine the relationship between levels of vitamin D and overall pulmonary function, as measured by PFTs (spirometry and body plethysmography).
  2. To determine effects of vitamin D supplementations on overall pulmonary function and selected biomarkers of inflammation (FeNO, pH, 8- isoprostane levels).
  Interventions: Drug: Vitamin D3
- Endocrine Arm (Experimental): Vitamin D3 Supplementation and Endocrine Function:
  To determine the effect of vitamin D replacement therapy on carbohydrate metabolism and insulin resistance in persons with vitamin D deficiency (<20ng/ml) and IGT, mild DM (e.g. fasting serum glucose <140 mg/dL) and/or IR.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 4000 IU/day or 2000 IU/day for 12 weeks
  Other Names: Cholecalciferol
  Arms: Endocrine Arm; Pulmonary Arm

SUMMARY:
Studies have shown that individuals who have suffered a spinal cord injury are at an increased risk of Vitamin D deficiency compared to able-bodied individuals. It has recently been shown that Vitamin D deficiency is linked to a large number of diseases and conditions, including chronic lung disease, vascular problems, and insulin resistance. If this common nutritional deficiency is proven to be the cause of some of these diseases and conditions in persons with SCI, then it may easily be remedied with a cheap and effective therapeutic approach: vitamin D replacement therapy. Because of the high prevalence of vitamin D deficiency in persons with SCI, this therapy alone or in combination with other treatment options will be expected to significantly improve overall well being in the SCI population, decrease hospitalization rate, and the lower the financial burden of care.

DETAILED DESCRIPTION:
Vitamin D deficiency is prevalent in individuals with Spinal Cord Injury (SCI). Recent studies have linked vitamin D with the prevention and/or treatment of a wide range of diseases, including chronic lung diseases. Patients with chronic lung diseases appear to be at increased risk for vitamin D deficiency for reasons that are not clear. Chronic lung diseases such as asthma and chronic obstructive lung disease (COPD) have been linked to vitamin D on a genetic basis. A recent observational study found a significant association between vitamin D deficiency and decreased pulmonary function in a large able-bodied population. The exact mechanisms involved have not been identified, but it has been postulated that vitamin D possesses a range of anti-inflammatory properties involving modulation of oxidative stress, or, possibly, protease/antiprotease balance and tissue damage/repair, mechanisms that have been shown to be important in the pathogenesis of chronic lung diseases. The relationship between vitamin D and the immune system is of utmost importance given that individuals with high cervical lesions express many obstructive aspects of pulmonary physiology commonly observed in individuals with asthma, in whom airway inflammation represents an underlying pathophysiological mechanism.

In addition to a high prevalence of vitamin D deficiency, persons with SCI have a higher prevalence of insulin resistance (IR), impaired glucose tolerance (IGT) and diabetes mellitus (DM). In the general population, vitamin D deficiency has been shown to be associated with IR, IGT and DM. If treatment of vitamin D deficiency in persons with SCI is shown to be associated with improvement in insulin sensitivity and reductions in impaired glucose tolerance or DM, then progression to more severe carbohydrate disorders may be delayed or prevented.

ELIGIBILITY:
Part 1: Screening for Vitamin D Deficiency

Inclusion Criteria:

* Between the ages of 18 and 75,
* Chronic (>1 year) SCI; tetraplegia (C3-8), paraplegia, (T1-6)

Exclusion Criteria:

* Acute illness
* Acute drug or alcohol use
* Lack of mental capacity to give informed consent,
* Pregnancy,
* Currently receiving Vitamin D supplementation.

Part 2A: Vitamin D and Pulmonary Function

Inclusion Criteria:

* Between the ages of 18 and 75,
* Chronic SCI (>1 year, C3-T6)
* Vitamin D deficiency as defined as a value <20 ng/ml.

Exclusion Criteria:

* Smoking, active or history of smoking during life time,
* Any history of blast injuries to the chest,
* Active respiratory disease,
* Pregnancy,
* Lack of mental capacity to give informed consent.
* Recent (within 3 months) respiratory infection.
* Receiving medications known to alter airway caliber.
* Acute drug or alcohol use,
* Currently receiving Vitamin D supplementation > 1000 units/day.

Part 2B: Vitamin D, Carbohydrate Metabolism, and Insulin Resistance

Inclusion Criteria:

* Between the ages of 18 and 75,
* Chronic SCI (>1 year, C3-T6)
* Vitamin D deficiency as defined as a value <20 ng/ml,
* Insulin Resistance (IR), Impaired glucose tolerance (IGT), and/or Diabetes Mellitus (DM).

Exclusion Criteria:

* Pregnancy,
* Problems with the kidneys,
* Lack of mental capacity to give informed consent,
* Acute drug or alcohol use,
* Currently receiving Vitamin D supplementation > 1000 units/day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of SCI participants with vitamin D deficiency | Screening study (1 visit, 2 hours)
  Vitamin D levels will be obtained during screening.

SECONDARY OUTCOMES:
Pulmonary function improvement as measured by PFTs in SCI with increased vitamin D levels | Change from baseline at 6 months
  Pulmonary function change will be measured in vitamin D deficient SCI subjects by spirometry and body plethysmography at baseline, 3 months, and 6 months.

OTHER OUTCOMES:
Pulmonary function improvement as measured by inflammation in SCI with vitamin D supplementation. | Change from baseline at 6 months
  Pulmonary function change will be measured in vitamin D deficient SCI subjects by biomarkers of inflammation, such as FeNO, pH, and 8-isoprostane, at baseline, 3 months, and 6 months.
Impaired glucose tolerance (IGT) improvement in SCI with vitamin D supplementation | Change from baseline at 6 months
  Vitamin D deficient SCI subjects with IGT and/or IR will undergo vitamin D replacement therapy. Glucose and insulin levels will be measured at baseline, 3 months, and 6 months.
Musculoskeletal pain improvement with vitamin D supplementation | Change from baseline at 6 months
  Vitamin D deficient SCI subjects will complete a pain survey at baseline, 3 months, and 6 months to assess musculoskeletal pain and how it may improve with vitamin D supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, M.D., Principal Investigator — James J Peters VA Medical Center
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided